CLINICAL TRIAL: NCT05221073
Title: Cross-cultural Adaptation and Psychometric Evaluation of the Bournemouth Questionnaire for Neck Pain
Brief Title: Urdu Version Of The Bournemouth Questionnaire For Neck Pain: A Reliability And Validity Study
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/FSD/0288
Record Dates: First submitted 2022-02-01; First posted 2022-02-02 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Neck Pain
Keywords: Bournemouth Questionnaire For Neck Pain; Neck Pain; Cultural adaptation; Validity; Urdu Version; Reliability
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of study is to translate & culturally adapt Neck Bournemouth Questionnaire into Urdu language along with investigation of the reliability & validity of Neck Bournemouth Questionnaire in General Population of Pakistan and to correlate with Neck Disability Index, Visual Analogue Scale, Neck Pain and Disability Scale and Rand 36-Item Health Survey

DETAILED DESCRIPTION:
The English version of the Bournemouth Questionnaire for Neck Pain will be translated and culturally adapted as per as previous recommendations. In the general population with neck pain, Urdu Version Of The Bournemouth Questionnaire For Neck Pain will be distributed among participants by choosing convenience sampling technique based on predefined inclusion and exclusion criteria. Test inter and intra- observer reliability of the final Urdu Version Of The Bournemouth Questionnaire For Neck Pain with Neck Disability Index, Neck Pain and Disability Scale, Visual Analogue Scale, and RAND will be filled with same day, by two observers and for the inter-observers assessment, with an interval of 45 minutes between the first and second application. Third assessment will be carried out after 7 days by Observer-1(re-intra-observers assessment. Data will be entered and analyzed by Cronbach alpha value. Test -retest reliability will be assessed using interclass correlation coefficient. The Urdu Version Of The Bournemouth Questionnaire For Neck Pain will be evaluated for content validity, construct validity, criterion validity and responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* 3 months of neck pain
* Neck pain more than six moth
* Male female both genders
* Physician referral
* Not prescribed medicine
* Without deformity in neck
* Ability of reading and writing

Exclusion Criteria:

* Joint inflammation or infection
* Pathology of shoulder
* Fibromylgia
* Psychologically unstable or having neurological disorder
* Cancer history
* Cervical injury
* Took treatment of physical therapy in last 6 month
* Any disability
* Loss of memory
* Disease or any Red flag
* Using Neck immobilization device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Population of Pakistan with Neck Pain was included in the study
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Neck Bournemouth Questionnaire | 1st day
  Neck Bournemouth Questionnaire contain seven dimensions tool used for the investigation of pain,functional ability, activity, depression,anxiety, work avoidance due to fear and control of pain
Neck Disability Index | 1st day
  The Neck Disability Index is most frequently used to evaluate pain in neck and neck pain related disability. One of previous study stated that the Neck Disability Index having multidisciplinary approach to disability
Visual Analogue Scale | 1st day
  Visual Analogue Scale provides a continuous scale for subjective magnitude estimation and consists of a straight line, the limits of which carry a verbal description of each extreme of the symptom to be evaluated. The line is usually 10 cm long and vertical, though different lengths and orientations have been employed and proven satisfactory.
Neck Pain and Disability Scale | 1st day
  The 20 items in the Neck Pain and Disability Scale measure the intensity of pain,its interference with the vocational,recreational,social, and functional aspects of living,and the presence and extent of associated emotional factors. The Neck Pain and Disability Scale is intended to be worded clearly and easy to complete.
Rand 36-Item Health Survey | 1st day
  Scoring the Rand 36-Item Health Survey 1.0 is a two-step process. First, preceded numeric values are recorded per the scoring key. Note that all items are scored so that a high score defines a more favourable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Ripah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No